CLINICAL TRIAL: NCT04831697
Title: Community-Based Intervention to Improve Diabetes Outcomes in Older African American Women With Multi-Caregiving Burden
Brief Title: Intervention to Improve Diabetes Outcomes in Older African American Women With Multi-Caregiving Burden
Acronym: MCGR21
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Joni Williams, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: R21DK123720 (NIH)
Record Dates: First submitted 2021-03-25; First posted 2021-04-05 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-Caregiving Intervention (Experimental): The multi-caregiving intervention consists of individual-based, social support, and health-educator facilitation and includes: a. Storytelling/sharing of experiences (5 minutes); social support and problem solving (15 minutes); Coping strategies (15minutes); and Structured Diabetes Education and Skills Training (15 minutes). The final 5min will be used for debriefing/reviewing goals.
  Interventions: Behavioral: Multi-Caregiving Intervention
- Diabetes Enhanced Usual Care Intervention (Active Comparator): This is composed of individual-based, health educator-facilitated diabetes education and skills training and general health education and will receive structured diabetes education and skills training as described above (30 minutes) and an additional discussion on general health topics (i.e., back pain, dyspepsia, etc.) (30 minutes).
  Interventions: Behavioral: Diabetes Enhanced Usual Care Intervention

INTERVENTIONS:
Behavioral: Multi-Caregiving Intervention — The multi-caregiving intervention consists of individual-based, social support, and health educator facilitation and includes: a. Storytelling/sharing of experiences (5 minutes); social support and problem solving (15 minutes); Coping strategies (15 minutes); and Structured Diabetes Education and Skills Training (15 minutes). The last 5 minutes will be used to debrief and review goals.
  Arms: Multi-Caregiving Intervention
Behavioral: Diabetes Enhanced Usual Care Intervention — This is composed of individual-based, health educator-facilitated diabetes education and skills training and general health education and will receive structured diabetes education and skills training as described above (30 minutes) and an additional discussion on general health topics (i.e., back pain, dyspepsia, etc.) (30 minutes).
  Arms: Diabetes Enhanced Usual Care Intervention

SUMMARY:
This is a two arm, pilot randomized control trial (RCT) in which 60 African American women (AAW), 40-64 years of age, with HbA1c ≥8% and multi-caregiving responsibilities will be recruited from communities in Milwaukee, Wisconsin and randomized to either: 1) an individual-based, social support, health educator-facilitated intervention to address multi-caregiving responsibilities (n=30), or 2) individual-based, health educator-facilitated diabetes education and skills training and general health education (n=30). All sessions will be delivered via telephone (i.e., landline, mobile device, smart device, etc.) by a health educator (i.e., nurse, social worker, Master's trained health educator) and is comprised of 12 weekly sessions and 3 booster sessions. Each session will last up to 60min. All study assessments will be administered by a Program Assistant at baseline, 3-months, and 6-months.

DETAILED DESCRIPTION:
The investigators propose to test the feasibility and preliminary efficacy of this multi-caregiving intervention on improving outcomes among AAW, ages 40-64 years with type 2 diabetes (T2DM) and multi-caregiving responsibilities using a pilot randomized design compared to diabetes enhanced usual care. The goals of the study will be assessed under the following specific aims:

Aim 1: To determine the feasibility of the multi-caregiving intervention as measured by recruitment, session attendance, retention, and treatment adherence in AAW with T2DM

Aim 2: To test the preliminary efficacy of the multi-caregiving intervention on glycemic and blood pressure control in AAW with T2DM compared to individual-delivered, health-educator led diabetes enhanced usual care at 6 months Hypothesis 1: AAW who receive the multi-caregiving intervention will have significant reductions in hemoglobin A1c at 6 months compared to AAW who receive diabetes enhanced usual care Hypothesis 2: AAW who receive the multi-caregiving intervention will have significant reductions in blood pressure at 6 months compared to AAW who receive diabetes enhanced usual care

Aim 3: To test the preliminary efficacy of the multi-caregiving intervention on self-care behaviors and quality of life in AAW with T2DM compared to individual-delivered, health educator led diabetes enhanced usual care at 6 months Hypothesis 1: AAW who receive the multi-caregiving intervention will have significant improvements in self-care behaviors (diet, physical activity, medication adherence, and blood glucose monitoring) at 6 months compared to AAW who receive diabetes enhanced usual care Hypothesis 2: AAW who receive the multi-caregiving intervention will have significant improvements in quality of life (SF-12 scores) at 6 months compared to AAW who receive diabetes enhanced usual care

In the final 6-month assessment, study participants will be asked to participate in 30 to 40-minute, semi-structured interviews by telephone. Findings will help refine the intervention and emphasize elements that enhance participant uptake and motivation for sustained behavior change for the future R01.

ELIGIBILITY:
Inclusion criteria:

* Age 40-64 years
* Self-identifies as female
* Self-identifies as African American or Non-Hispanic Black
* Self-reports multi-caregiving responsibilities
* Clinical diagnosis of T2DM based on HbA1c≥8% at the screening/baseline assessment
* Able to communicate in English
* Access to a telephone (i.e., landline, mobile device, smart device, etc.)

Exclusion criteria:

* Mental confusion at screening/baseline assessment suggesting significant dementia, active psychosis, or acute mental disorder
* Participation in other diabetes trials
* Life expectancy <6 months based on screening questionnaire

Ages: 40 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Glycemic Control from Baseline to 6 months | Screening/Baseline, 3-months, 6-months
  Trained personnel will collect a blood specimen via finger stick (using a Point-of-Care device) or via venipuncture to collect 10cc of blood to measure HbA1c. All collections will be performed in the community at a location convenient to the study participant. At the screening visit, the HbA1c must be 8% or greater to be eligible for participation.

SECONDARY OUTCOMES:
Change in Diet from Baseline to 6 months | Screening/Baseline, 3-months, 6-months
  Diet will be measured by the 26-item Dietary Screener Questionnaire (DSQ) used in the National Health and Nutrition Examination Survey. Responses are used to estimate individual dietary intake for fruits, vegetables, dairy, added sugars, whole grains, fiber, adn calcium.
Change in Physical Activity from Baseline to 6 months | Screening/Baseline, 3-months, 6-months
  Physical activity will be measured using the 7-item International Physical Activity Questionnaire that asks about physical activities over the last 7 days.
Change in Blood Pressure Control from Baseline to 6 months | Screening/Baseline, 3-months, 6-months
  Blood pressure measurements will be obtained by the nurse/health educator using an automated BP monitor with participants seated comfortably for 5 minutes prior to the measurements.
Change in Blood Glucose Monitoring from Baseline to 6 months | Screening/Baseline, 3-months, 6-months
  Blood glucose monitoring will be assessed with the previously validated Summary of Diabetes Self-Care Activities (SDSCA) scale, where scores are calculated for each of the five areas assessed by the SDSCA over the past 7 days: diet, exercise, blood glucose monitoring, foot care, and smoking status. Higher scores mean more engagement in self-care behaviors.
Change in Medication Adherence from Baseline to 6 months | Screening/Baseline, 3-months, 6-months
  Medication adherence will be measured with the 6-item validated self-report Brooks Medication Adherence Scale. Each question asks yes-no questions about adherence, where a "no" response indicates better adherence.
Change in Health Related Quality of Life from Baseline to 6 months | Screening/Baseline, 3-months, 6-months
  The SF-12 is a valid and reliable instrument to measure functional status and yields summary physical (PCS-12) and mental health (MCS-12) outcome scores. Summary scores range from 0 to 100 where higher scores mean better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Joni Williams, MD, MPH, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States